CLINICAL TRIAL: NCT00452283
Title: The Effect of a Systemic Non-selective Endothelin Antagonist on Intraocular Pressure and Anterior Depth in Pulmonary Hypertension Patients.
Brief Title: Changes in Eye Pressure and Anterior Chamber Depth With Oral Endothelin Antagonist Therapy
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 06-0792
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Glaucoma; Pulmonary Hypertension
MeSH Terms: conditions — Glaucoma; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is growing evidence that a cause of glaucoma is linked to circulatory problems and poor auto-regulation of blood flow to the optic nerve. Pulmonary hypertension (PH)is a disease characterized by low oxygen levels in the blood and altered blood circulation. The decrease in oxygen delivery to the optic nerve could lead to the loss of nerve fiber layer(NFL)in the retina and the resulting visual field compromise. This situation is characteristic of glaucoma. The ability to identify NFL thinning early could lead to earlier diagnosis of glaucoma and more effective treatment to limit dysfunction from visual field loss.

We hypothesize that the rate of structural damage to the NFL, a feature of glaucoma, is higher in patients with PH than expected in healthy populations lacking this disease.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with pulmonary hypertension
* between the ages of 18 and 80 years
* ability to undergo the various ocular exams.

Exclusion Criteria:

* patients with other diseases that could affect the nerve fiber layer
* special populations; ie children, pregnancy, lactating females, prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2007-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Occurence of nerve fiber layer abnormalities | Single Exam

SECONDARY OUTCOMES:
Optic Nerve Head Structure | Single Exam

OTHER OUTCOMES:
Visual Field Defects | Single Exam
Retinal Blood Flow Changes | Single Exam

CONTACTS AND LOCATIONS:
Overall Officials: Malik Y. Kahook, M.D., Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Eye Center, Aurora, Colorado, United States